CLINICAL TRIAL: NCT05501535
Title: Objective Refraction Changes After Using ND: YAG LASER In Treatment of Posterior Capsular Opacification In Pseudo Phakic Eye After Successful Non Complicated Cataract Surgery
Brief Title: Refraction Changes After Using ND: YAG LASER In Treatment of Posterior Capsular Opacification In Pseudo Phakic Eye
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Mohmamed Elsayed Mohamed Ahmed, Principal investigator, Sohag University
Other Study IDs: Soh-Med-22-08-05
Record Dates: First submitted 2022-08-11; First posted 2022-08-15 (Actual); Last update posted 2022-08-17 (Actual); Status verified 2022-08

CONDITIONS: Posterior Capsule Opacification

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Device: Yes

GROUPS / COHORTS (1):
- pseudophakic patients before and after having ND YAG laser
  Interventions: Device: ND:YAG LASER

INTERVENTIONS:
Device: ND:YAG LASER — The standard therapy for PCO is now Nd: YAG laser posterior capsulotomy, which has a success rate of more than 95%. The neodymium: yttrium-aluminum-garnet (Nd:YAG) laser, with a wavelength of 1064 nm, is a solid-state laser that may destroy ocular tissues by achieving optical breakdown with a brief, high-power pulse .Ionization or plasma production occurs in the ocular tissue as a result of optical breakdown. This plasma production subsequently generates acoustic and shock waves, which destroy tissue. Because of its cost-effectiveness, speed, and lack of invasiveness, it is the chosen treatment option in PCO

SUMMARY:
The most prevalent long term consequence of cataract surgery in both phacoemulsification and extracapsular cataract excision is posterior capsular opacification (PCO) PCO occurred in 11.8 percent of patients one year after surgery, 20.7 percent in three years, and 28.4 percent in five years .

It causes lower visual acuity, decreased contrast sensitivity, stereoscopic vision, increases glare and monocular diplopia. The pathogenesis of PCO is dependent on the growth of lens epithelial cell remnants in the intracapsular region. Continuous curvilinear capsulorhexis, good hydro dissection, efficient removal of cortical and lenticular epithelial cells, in-the-bag IOL implantation, and the use of single-piece acrylic sharp edges IOLs are all factors in PCO avoidance. Intraoperatively, anti-metabolites such as 5-fluorouracil and mitomycin C may also be utilized.

Fortunately, the overall prevalence of PCO and the using of neodymium-yttrium-aluminum-garnet (Nd: YAG) laser posterior Capsulotomy rates have dropped from 50% to fewer than 10% now The standard therapy for PCO is now Nd: YAG laser posterior capsulotomy, which has a success rate of more than 95%. The neodymium: yttrium-aluminum-garnet (Nd:YAG) laser, with a wavelength of 1064 nm, is a solid-state laser that may destroy ocular tissues by achieving optical breakdown with a brief, high-power pulse .Ionization or plasma production occurs in the ocular tissue as a result of optical breakdown. This plasma production subsequently generates acoustic and shock waves, which destroy tissue. Because of its cost-effectiveness, speed, and lack of invasiveness, it is the chosen treatment option in PCO.

However laser capsulotomy is not free of complications including transient intraocular pressure (IOP) elevation, hyphema, uveitis, cystoid macular edema, and retinal detachments that occur most frequently in the first few months . Apart from the afore mentioned biological complications, mechanical effects of laser capsulotomy such as pitting of IOL, dislocation of IOL into the vitreous, and shift in the position of IOL have also be reported Displacement of the IOL following laser capsulotomy, which may be impacted by the capsulotomy size , might hypothetically modify the effective power of the IOL as well as the patients' refractive state may be altered . However, with the exception of one research that demonstrated a hyperopic shift after Nd:YAG laser capsulotomy , most prior investigations failed to show a significant change in refraction before and after Nd:YAG laser capsulotomy . According to earlier study , the size and form of Nd:YAG laser capsulotomy, the energy utilized in Nd:YAG laser capsulotomy, and the designs of IOL did not alter the post-laser refractive state.

It is still unknown if the time of laser capsulotomy affects the refractive and visual prognosis of patients after Nd:YAG laser capsulotomy. Because the IOL would continue to rotate for at least 6 months following cataract surgery, Any considerable change in IOL position might result in a change in the patient's refractive state, necessitating corrective lens prescriptions

ELIGIBILITY:
Inclusion Criteria :

• presence of clinically significant central Posterior capsular opacification

Exclusion Criteria:

* High Intra ocular pressure
* Corneal opacities or dystrophies.
* Dense posterior capsular opacification where no refraction could be obtained

Ages: 40 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: sohag university hospital patients in ophthalmology clinc
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-11-01 (Estimated)

PRIMARY OUTCOMES:
objective refractive changes in sphere and cylinder refraction | one month
  using autorefractometer

CONTACTS AND LOCATIONS:
Overall Officials: mohamed elagouz, prof, Study Chair — unaffilatted
Locations (1):
- Sohag university hospital, Sohag, Egypt

IPD SHARING:
Plan to Share IPD: Yes
All patients will be evaluated eventually one month after the procedure which included BCVA and slit lamp examination. Patients undergo retinoscopy and auto-refractometer . Then subjective refraction will be performed and readings will be documented. The changes in refraction will be noted and analyzed. Spherical and cylindrical error shift post procedure will be determined The collected data will be tabulated, coded and analyzed using SPSS program,
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 months after publication